CLINICAL TRIAL: NCT04272177
Title: Influence of Shared-Decision Making in Reducing Decision Conflict on the Choice of Awakening Agent After General Anesthesia: A Multicenter Randomized Controlled Trial
Brief Title: Influence of Shared-Decision Making in Reducing Decision Conflict on the Choice of Awakening Agent After General Anesthesia
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Taipei Medical University Shuang Ho Hospital (Other)
Collaborators: Chi Mei Medical Hospital (Other)
Responsible Party: Principal Investigator, Ka-Wai Tam, Director of Shared Decision Making Resource Center, Taipei Medical University Shuang Ho Hospital
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Health Services Research
Other Study IDs: N201909073; 10812-015 (Other: Chi Mei Medical Center)
Record Dates: First submitted 2020-02-13; First posted 2020-02-17 (Actual); Last update posted 2021-03-19 (Actual); Status verified 2021-03

CONDITIONS: Decision Making, Shared
Keywords: shared decision making, sugammadex, patient decision aids

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- SDM group (Experimental): Shared decision making using PDAs. PDAs is used as a tool explain the advantages and disadvantages of the traditional reversal drugs and sugammadex. And by following SDM principles, the patients are guided to consider their individual values and preferences and helped to make a choice that best meet their needs.
  Interventions: Other: Shared decision making with the used of patient decision aids
- Control group (No Intervention): Current approach to explain details of anesthesia using a single introductory sheet made by the two hospitals or provided by the pharmaceutical companies is used.

INTERVENTIONS:
Other: Shared decision making with the used of patient decision aids — PDA is used to explain choices of reversal drugs using SDM approach during consultation. The patients and medical staff explore the preferences with PDA and make decision together.
  Arms: SDM group

SUMMARY:
General anesthesia is an important procedure for patients undergoing a surgery. When awakening is required after the surgery, the supply of anesthetic gas is terminated together with the administration of reversal drugs. Acetylcholinesterase inhibitors were the main drugs of choice in the past, most of the patients will awake in 15 to 30 minutes. The breathing circuit will then be extracted when patient breathing has recovered to normal.

sugammadex, a new generation reversal drug, is a type of selective relaxant-binding agent which recover patient muscle and breathing activities at around 3 minutes. In comparison with neostigmine, sugammadex has a shorter awakening time and lower risk of bradycardia, postoperative nausea vomiting, and postoperative residual paralysis. However, the drug has not been widely applied in Taiwan because it is not covered by the national insurance. We believe it would the patients to understand the characteristics of sugammadex in fair perspectives and increase the operation power of surgical rooms if shared decision making with the use of Patient Decision Aids (PDAs) is used during anesthesia consultation.

DETAILED DESCRIPTION:
Background:

A PDA was developed to be administered during anethesia consultation for surgical patients. We expect the PDA would benefit the intervention group in the aspects of knowledge and communication in choosing reversal drugs.The aim of this study is to conduct a multicenter randomized controlled trial (RCT) to evaluate the benefit of PDAs on decision making.

Patients and Methods:

Decision aids are interventions designed to help surgical patients with general anethesia to choose their options of neostigmine or sugammadex by providing information on those options. In this multicenter RCT, surgical patients are randomly divided into SDM and control groups. In control group, patients will receive details of anesthesia using single introductory sheet. In SDM group, PDA will be used as a tool to explain the benefits and harms between the traditional reversal drugs and sugammadex. And by following SDM principles, the patients are guided to consider their individual values and preferences and helped to make a choice that best meet their needs. This study will be conducted in 2 hospitals (Shuang Ho Hospital and Chi Mei Medical Center). The outcomes are decision conflicts and decision-making difficulties after consultation of the patients.

Hypothesis:

The patients of the SDM group are predicted to have lower decisional conflict scores and higher knowledge scores when compared with controlled group. Our study hopes to support the efficacy of PDAs in helping surgical patients to make a choice that best meet their needs.

ELIGIBILITY:
Inclusion Criteria:

1. Patients who receive general anesthesia
2. Adults older than 20 years
3. Communicable with Mandarin
4. Patients who receive anesthesia consulting

Exclusion Criteria:

1. Patients who do not receive general anesthesia
2. Patients receive spinal anesthesia
3. Not communicable with Mandarin.
4. Emergency patient who do not receive anesthesia consulting

Ages: 20 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 3309 (Actual)
Dates: Start 2020-03-20 (Actual); Primary Completion 2020-08-20 (Actual); Study Completion 2020-09-20 (Actual)

PRIMARY OUTCOMES:
Decision conflicts | One day after surgery
  Mean score of decisional conflict scale by SURE test (developed by Ottawa University) using a five-item scale: 1. disagree strongly; 2. disagree; 3. neutral; 4. agree; 5. agree strongly.
Knowledge | One day after surgery
  Mean score of understanding of reversal drugs by SURE test (developed by Ottawa University) using a five-item scale: 1. disagree strongly; 2. disagree; 3. neutral; 4. agree; 5. agree strongly.

SECONDARY OUTCOMES:
Percentage of choices of reversal drugs | 10 minutes before anesthesia
  Percentage of choices of reversal drugs

CONTACTS AND LOCATIONS:
Locations (1):
- Shuang Ho Hospital, Taipei Medical University, New Taipei City, Taiwan

IPD SHARING:
Plan to Share IPD: Yes